CLINICAL TRIAL: NCT01890356
Title: A Study of Transcranial Electrical Stimulation (TES) as a Maintenance Treatment for Depression
Brief Title: Maintenance Transcranial Electrical Stimulation for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Colleen Loo, Professor, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HC12499
Record Dates: First submitted 2013-06-26; First posted 2013-07-01 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder; Bipolar Disorder
Keywords: Depression; Treatment; Transcranial electrical stimulation; Maintenance
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Depression | interventions — Transcranial Direct Current Stimulation

ARMS (1):
- Transcranial electrical stimulation (Experimental)
  Interventions: Device: Transcranial electrical stimulation

INTERVENTIONS:
Device: Transcranial electrical stimulation

SUMMARY:
Transcranial electrical stimulation (TES) techniques offer a novel treatment approach for depression and have shown promising efficacy. However, there is no published data to date on their effectiveness as a maintenance treatment. This study will investigate ways of using TES as a maintenance treatment to prevent relapse in depression.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be ≥ 18 years old.
* Participants must have experienced a significant clinical response, defined as ≥ 50% decrease from baseline scores on the Montgomery Asberg Depression Rating Scale (MADRS).

Exclusion Criteria:

* Inadequate response to acute trial of TES.
* Suicidality.
* Clinically defined neurological disorder or insult.
* Metal in the cranium, skull defects, or skin lesions on scalp (cuts, abrasions, rash) at proposed electrode sites.
* Pregnancy (women of childbearing age will be asked to undergo a urine pregnancy test prior to starting the study).
* Concurrent long acting benzodiazepines, ritalin or dexamphetamine medication.
* Treatment for depression is changed during months 3-9 of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-06; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale for Depression (MADRS) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Loo, MBBS, Principal Investigator — University of New South Wales
Locations (1):
- Black Dog Institute / University of New South Wales, Randwick, Sydney, New South Wales, Australia